CLINICAL TRIAL: NCT00736996
Title: Pioglitazone and Exercise Effects on Older Adults With MCI and Metabolic Syndrome
Brief Title: Pioglitazone Or Exercise to Treat Mild Cognitive Impairment (MCI)
Acronym: POEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-1215; R01AG028746 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Metabolic Syndrome; Mild Cognitive Impairment; Insulin Resistance; Endurance Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Metabolic Syndrome; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pioglitazone (Experimental): Pioglitazone
  30 - 45mg tablet daily for 6 months
  Interventions: Drug: Pioglitazone
- Endurance Exercise Training (Active Comparator): Endurance Exercise Training (EET) Individualized exercise prescription, 45-75 minutes (progressive increments) three times a week
  Interventions: Behavioral: Endurance Exercise Training
- Placebo (Placebo Comparator): Placebo matching tablet sugar pill daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 30 - 45mg tablet daily for 6 months
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Matching tablet daily for 6 months
  Arms: Placebo
Behavioral: Endurance Exercise Training — Individualized exercise prescription, 45-75 minutes (progressive increments) three times a week
  Arms: Endurance Exercise Training

SUMMARY:
The purpose of this study is to investigate novel treatments to delay progression to dementia in patients with mild cognitive impairment (MCI) and metabolic syndrome (MS). The hypothesis is that treatment with pioglitazone or endurance exercise training will improve, stabilize, or attenuate decline in cognitive function compared to controls. This study will also discover potential mechanisms for the improvements and determine the baseline prevalence of amnestic versus non-amnestic MCI.

DETAILED DESCRIPTION:
The Metabolic Syndrome (MS) is a rapidly growing public health problem. This constellation of metabolic abnormalities increases the risk of diabetes, heart disease and death. Recently evidence has linked MS with cognitive impairment and dementia, including Alzheimer's Disease (AD). AD is preceded by a state called Mild Cognitive Impairment (MCI), characterized by subjective and objective memory impairment, but no functional impairment. Although not all persons with MCI will develop AD, the conversion rate from MCI to AD is about 15% per year, or 5-10 times that of cognitively normal individuals. There is great interest in finding treatments to prevent AD by intervening at an earlier stage, i.e. MCI.

The mechanism(s) linking MS and cognitive impairment are not clear, although there is evidence that insulin resistance and inflammation play key roles. Thiazolidinediones (TZDs) are medications approved for the treatment of Type 2 Diabetes, which work by reducing insulin resistance. In addition, these drugs have anti-inflammatory properties. A recent pilot study showed improvements in some areas of cognition in patients with MCI or mild AD treated with the TZD rosiglitazone. Endurance exercise training (EET) is an established treatment for MS and insulin resistance. There is also evidence that EET may improve cognitive function as well.

Adults aged 55 years or older with both MS and MCI at baseline will be randomized to a 6-month intervention with either (1) treatment with pioglitazone, (2) endurance exercise training, or (3) control (placebo and no exercise). The hypothesis is that treatment with the TZD pioglitazone or EET will improve cognitive function compared to controls, as evidenced by either improvement, stabilization, or lesser decline in performance on cognitive testing. Participants will undergo a physical exam including blood and urine tests, a complete neurologic exam, and a comprehensive battery of cognitive tests. They will also have a DEXA scan, exercise treadmill test, non-invasive tests of vascular function and a hyperglycemic-euglycemic clamp procedure to measure insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling, over 55 years old, able to give full informed consent, willing to be randomized
* Able to perform a telephone interview
* Able to speak, read and understand English
* Potential volunteers on a statin drug, angiotensin converting enzyme inhibitor (ACE-I), angiotensin II receptor blocker (ARB), non-steroidal anti-inflammatory drug (NSAID), or Vitamin E supplement, are eligible but must be on a stable dose for at least 2 months
* Women must be post-menopausal, as defined by no menses for 12 months
* Must meet 3 of the 5 requirements for Metabolic Syndrome:

  * Waist measurement: greater than 102 cm for men and 88 cm for women
  * Fasting hypertriglyceridemia: 150 mg/dl (1.7 mmol/L) or higher
  * Low HDL cholesterol: less than 40 mg/dl (1.0 mmol/L) for men and 50 mg/dl (1.3 mmol/L) for women
  * Hypertension: higher than 130 mmHg systolic or 85 mmHg diastolic (average of 2 seated measurements) or currently using an antihypertensive medication
  * Elevated (untreated) fasting glucose: 100 mg/dl (5.6 mmol/L) or higher
* Meet the study's 4-step screening process for MCI (to rule out dementia)

Exclusion Criteria:

* Diagnosis of diabetes mellitus (DM), defined as: Fasting Blood Sugar 126 or higher, a history of known DM, or treatment with any glucose lowering medication
* Current diagnosis of dementia (or MMSE less than 24) or a neurological co-morbidity other than MCI that might affect cognition including: large vessel stroke, brain tumor, severe brain injury, multiple sclerosis, or Parkinson's disease
* Current diagnosis of depression assessed by a Centers for Epidemiologic Studies Depression Scale (CES-D) score of 36 or less
* Major psychiatric conditions such as bipolar disorder, psychosis, schizophrenia, or alcoholism that could affect the ability to understand and/or cooperate fully with the protocol
* Significant cerebral vascular disease
* Modified Hachinski score greater than 4
* Pregnant, lactating or having child bearing potential
* Concomitant medications with significant cholinergic or anticholinergic effects or adverse effects on cognition including: antipsychotics, tricyclic antidepressants, anticonvulsants, sedative/hypnotics, anxiolytics, glucocorticoids (chronic or frequent intermittent), gingko biloba, NMDA receptor antagonists, cholinesterase inhibitors, strongly lipid soluble beta blockers (e.g., propranolol)
* Hormone replacement therapy (male or female)
* Visual/hearing impairment that would significantly impact the ability to undergo psychometric testing
* Significant medical illness or organ failure including hepatic or renal failure, unstable cardiac disease, or life expectancy less than 18 months
* Exercise-limiting conditions including: neuromuscular, joint/bone, cardiovascular, peripheral vascular, cerebrovascular or pulmonary disease; recent MI, pulmonary embolus, significant aortic stenosis; or exercise limiting obesity
* Untreated B12 deficiency or hypothyroidism (stable treatment for at least 3 months is allowable)
* Uncontrolled hypertension: over 160 mmHg systolic or 100 mmHg diastolic (stable treatment is allowable)
* Endurance exercise training more than twice a week for 20 minutes (at a level that produces sweating) consistently during the last 6 months
* Unstable weight in the last 6 months
* Increased risk for Pio toxicity including: a) baseline liver dysfunction (over 2.5xULN for AST, ALT); b) hematocrit less than 33% men or 30% women; c) problematic edema; or d) congestive heart failure NYHA class II or greater
* Stage 5 renal impairment (GFR less than 15 or dialysis)
* Already taking a TZD or other drug that would modify insulin resistance (e.g. metformin), or has taken a TZD in the past and experienced a significant adverse effect or allergy
* Currently taking any of following medications that may interact with Pio metabolism: atorvastatin at 80mg/day (lower doses are allowed), and medications with major CYP 3A4 inhibiting effects, such as nefazodone or systemic antifungal agents
* Participating in another clinical trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Schwartz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Denver, Colorado, United States

REFERENCES:
- [Background] Kramer AF, Erickson KI, Colcombe SJ. Exercise, cognition, and the aging brain. J Appl Physiol (1985). 2006 Oct;101(4):1237-42. doi: 10.1152/japplphysiol.00500.2006. Epub 2006 Jun 15. PMID 16778001
- [Background] Yaffe K, Kanaya A, Lindquist K, Simonsick EM, Harris T, Shorr RI, Tylavsky FA, Newman AB. The metabolic syndrome, inflammation, and risk of cognitive decline. JAMA. 2004 Nov 10;292(18):2237-42. doi: 10.1001/jama.292.18.2237. PMID 15536110
- [Background] Steen E, Terry BM, Rivera EJ, Cannon JL, Neely TR, Tavares R, Xu XJ, Wands JR, de la Monte SM. Impaired insulin and insulin-like growth factor expression and signaling mechanisms in Alzheimer's disease--is this type 3 diabetes? J Alzheimers Dis. 2005 Feb;7(1):63-80. doi: 10.3233/jad-2005-7107. PMID 15750215
- [Background] Watson GS, Cholerton BA, Reger MA, Baker LD, Plymate SR, Asthana S, Fishel MA, Kulstad JJ, Green PS, Cook DG, Kahn SE, Keeling ML, Craft S. Preserved cognition in patients with early Alzheimer disease and amnestic mild cognitive impairment during treatment with rosiglitazone: a preliminary study. Am J Geriatr Psychiatry. 2005 Nov;13(11):950-8. doi: 10.1176/appi.ajgp.13.11.950. PMID 16286438
- [Background] Lytle ME, Vander Bilt J, Pandav RS, Dodge HH, Ganguli M. Exercise level and cognitive decline: the MoVIES project. Alzheimer Dis Assoc Disord. 2004 Apr-Jun;18(2):57-64. doi: 10.1097/01.wad.0000126614.87955.79. PMID 15249848

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone: Pioglitazone: 45mg oral tablet daily for 6 months
- Endurance Exercise Training: Endurance Exercise Training: Supervised, thrice-weekly, 45-75 minute sessions of treadmill walking, initially moderate intensity (50-60% of maximum heart rate), with progressive increases in intensity to the best of the subject's ability, up to 85% of maximal heart rate.
- Placebo: Placebo: Matching oral tablet daily for 6 months
Period: Overall Study
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo
Started | 25 | 26 | 27
Completed | 24 | 17 | 25
Not Completed | 1 | 9 | 2
Not completed — Lost to Follow-up | 1 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo | Total
Number analyzed (Participants) | 24 | 17 | 25 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6) | 64 (7) | 68 (7) | 65 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 15 | 35
  Male | 11 | 10 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 0 | 4
  Not Hispanic or Latino | 20 | 17 | 24 | 61
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 20 | 15 | 23 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 17 | 25 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Performance
Description: Participants were administered a neuropsychological testing battery consisting of assessments in four cognitive domains: memory (Visual Reproduction II, Logical Memory II, Rey Auditory Verbal Learning Test), language (Boston Naming Test , Category Fluency), visuospatial (Block Design, Picture Completion), and executive function (Trail Making Test B, Digit Symbol Test). Raw test scores for these primary cognitive domain measures were transformed into age-adjusted scaled scores with a mean of 10 and a standard deviation (SD) of 3, with higher numbers indicating better cognitive performance, using the Mayo's Older American Normative Studies data. Cognitive domain scores were calculated as the arithmetic mean of the normatively derived scaled scores for all of the tests in that domain.
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo
Number analyzed (Participants) | 24 | 17 | 25
units on a scale
  Memory domain | 0.8 [-1.4 to 2.9] | 0.7 [-1.5 to 2.8] | 1.2 [-1.0 to 3.4]
  Language domain | 0.4 [-1.8 to 2.6] | 0.6 [-1.6 to 2.8] | 0.4 [-1.9 to 2.6]
  Visuospatial domain | 0.3 [-1.7 to 2.3] | 1.1 [-0.9 to 3.1] | 0.8 [-1.2 to 2.8]
  Executive function domain | 1.0 [-0.9 to 3.0] | 0.7 [-1.2 to 2.6] | 0.9 [-1.1 to 2.9]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; The mean change in domain score with PIO was compared with the mean change in domain score with Placebo in a linear regression conditioned on the stratification categories (MCI subtype and number of APOE ε4 alleles) and the baseline domain score; Test type: Superiority or Other; p < 0.0125, Regression, Linear — Statistical significance was defined as a 2-sided p-value < 0.0125 (=0.05/4) to adjust for multiple comparisons
Statistical Analysis 2: Comparison: Endurance Exercise Training vs Placebo; The mean change in domain score with EET was compared with the mean change in domain score with Placebo in a linear regression conditioned on the stratification categories (MCI subtype and number of APOE ε4 alleles) and the baseline domain score; Test type: Superiority or Other; p < 0.0125, Regression, Linear — Statistical significance was defined as a 2-sided p-value < 0.0125 (=0.05/4) to adjust for multiple comparisons

2. Secondary Outcome: Change in Insulin Resistance
Description: Change in whole body glucose disposal rate (mg/kg/min) calculated during a single-stage (40 mU/m2/min), 3-hour hyperinsulinemic, euglycemic clamp
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: mg/kg/min
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo
Number analyzed (Participants) | 24 | 17 | 25
mg/kg/min | 1.7 [0.9 to 2.4] | 0.7 [-0.1 to 1.6] | 0.1 [-0.6 to 0.8]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; The mean change with PIO was compared with the mean change with Placebo in a linear regression conditioned on the stratification categories (MCI subtype and number of APOE ε4 alleles) and the baseline level of the outcome variable; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Endurance Exercise Training vs Placebo; The mean change with EET was compared with the mean change with Placebo in a linear regression conditioned on the stratification categories (MCI subtype and number of APOE ε4 alleles) and the baseline level of the outcome variable; Test type: Superiority or Other; p < 0.05, Regression, Linear

3. Secondary Outcome: Change in Peak Oxygen Uptake (VO2 Peak)
Description: Peak oxygen consumption (VO2 peak, ml/kg/min) was determined by open circuit spirometry during a standard treadmill stress test (modified Balke protocol).
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo
Number analyzed (Participants) | 24 | 17 | 25
ml/kg/min | 0.9 [-4.6 to 6.4] | 3.2 [-2.3 to 8.7] | 1.3 [-4.1 to 6.7]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Endurance Exercise Training vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pioglitazone | Endurance Exercise Training | Placebo
Serious Adverse Events (participants affected / at risk) | 3/25 | 1/26 | 3/27
Other Adverse Events (participants affected / at risk) | 18/25 | 19/26 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=25) | Endurance Exercise Training (N=26) | Placebo (N=27)
Paroxysmal supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Incorrect insulin dosage infused during clamp study
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Kidney mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=25) | Endurance Exercise Training (N=26) | Placebo (N=27)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (4) | 11 (11) | 6 (6)
Cardiovascular (Cardiac disorders) | 4 (5) | 2 (2) | 4 (5) — Includes lower extremity edema
Dermatologic (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 5 (5)
Gastrointestinal (Gastrointestinal disorders) | 5 (6) | 6 (7) | 4 (4)
General (General disorders) | 10 (10) | 5 (8) | 6 (6)
ENT (Ear and labyrinth disorders) | 3 (4) | 1 (1) | 1 (1)
Endocrine (Endocrine disorders) | 0 (0) | 3 (5) | 1 (2)
Hematologic (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Genitourinary (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (4)
Neurologic (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Behavioral (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Infectious Disease (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Opthalmologic (Eye disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No